CLINICAL TRIAL: NCT06496893
Title: A Randomized, Double-blind, Placebo-controlled Study to Assess the Effect of Glucocil® on Metabolic Health in Individuals With Prediabetes and Type 2 Diabetes Mellitus.
Brief Title: A Study to Assess Effect of Glucocil® on Metabolic Health in Individuals With Prediabetes and Type 2 Diabetes Mellitus.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NH/231201/GC/DM
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Pre Diabetes; Type2 Diabetes Mellitus
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active 1200 mg per soft gel capsule (Active Comparator): Combination of Vitamin B1, B6, B12, D3, Chromium Picolinate, Proprietary Mulberry Leaf Extract, Cinnamon Bark Powder, Gymnema Sylvestre Extract, Insulina (Cissus Sicyoides) Leaf Extract, Alpha Lipoic Acid, Phellodendron Bark Extract (Berberine HCL), Cissus Quadrangularis Extract, Banaba Leaf Extract, & Fish Oil.
  Two soft gels to be taken with breakfast and two soft gels to be taken with dinner
  Interventions: Dietary Supplement: IP 1200 mg per soft gel capsule
- Placebo (Soyabean oil) 1200 mg per soft gel capsule (Placebo Comparator): Two soft gels to be taken with breakfast and two soft gels to be taken with dinner
  Interventions: Dietary Supplement: Placebo Comparator: Placebo 1200 mg per soft gel capsule

INTERVENTIONS:
Dietary Supplement: IP 1200 mg per soft gel capsule — Two soft gels to be taken with breakfast and two soft gels to be taken with dinner
  Arms: Active 1200 mg per soft gel capsule
Dietary Supplement: Placebo Comparator: Placebo 1200 mg per soft gel capsule — Two soft gels to be taken with breakfast and two soft gels to be taken with dinner
  Arms: Placebo (Soyabean oil) 1200 mg per soft gel capsule

SUMMARY:
A randomized, double-blind, placebo-controlled study to assess the effect of Glucocil® on metabolic health in individuals with prediabetes and Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study to assess the effect of Glucocil® on metabolic health in individuals with prediabetes and Type 2 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of age more than equal to 30 years and less than equal to 70 years.
2. Body mass index within 30 kg/m2 and 35 kg/m2 (both values included) with waist circumference above 40 inches (men) or 35 inches (women).
3. Cohort 1 (Only for prediabetes individuals)- Individuals diagnosed with prediabetes with OGTT (140 mg/dL to 199 mg/dL); HbA1c (5.7% to 6.9%) and fasting blood glucose level (between 100 mg/dL to 125 mg/dL).
4. Cohort 2 (T2DM)- Individuals newly diagnosed with Type 2 diabetes mellitus with HbA1c between 7% and 9% (both values included) and fasting blood glucose level in between 126 to 180 mg/dL.
5. Triglycerides between 150 mg/dL and 299 mg/dL (both values inclusive) and/or Low-Density Lipoprotein (LDL) in between 130 mg/dL and 189 mg/dL (both values inclusive).
6. Individuals having non-vegetarian diet for at least 2 days a week.
7. Non-smoker.
8. Individuals who are willing to not change their physical activity levels throughout the study period.
9. Individuals willing to complete all study-related questionnaires and to complete all clinical study visits.
10. Individuals ready to give voluntary, written informed consent to participate in the study.

Exclusion Criteria:

1. Individuals who are exclusively vegetarians diet.
2. Individuals with Type 1 diabetes mellitus.
3. Individuals with Type 2 diabetes mellitus on medication.
4. Individuals with any other endocrine disorder.
5. Individuals who are currently on diuretics or thyroid supplements
6. Individuals on lipid-lowering therapies.
7. Individuals with uncontrolled hypertenstion as assessed by systolic over diastolic blood pressure (≥ 140/90 mmHg).
8. Individuals who are currently on antihypertensive medication.
9. Individuals with cardiac arrhythmia, impaired hepatic or renal function
10. Individuals having heart failure, coronary artery disease, hyperthyroidism, hypothyroidism, cancer or mental disease or any other serious disease requiring active treatment.
11. History of malignancy or stroke.
12. Chronic alcoholism: History and/or current cases of chronic alcohol consumption or heavy drinkers as defined by i.For men consuming more than 4 drinks on any day or more than 14 drinks/week ii. For women, consuming more than 3 drinks on any day or more than 7 drinks/week
13. Individuals taking concomitant medication known to alter blood sugar.
14. Individuals having treatment with herbal or any other supplements.
15. Any condition or abnormality that would compromise the safety of the individuals or the quality of the study data.
16. Use of another investigational product within 3 months of the screening visit.
17. Females who are lactating, pregnant or planning to be pregnant or taking any oral contraceptives

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 2- (Type 2 diabetes mellitus (T2DM)) To assess the effect of Investigational Product (IP) on blood sugar as assessed by Glycated haemoglobin (HbA1c) in individuals with Type 2 diabetes mellitus (T2DM). | Screening visit (The same value will be considered for baseline) and Day 90.
  HbA1c reference ranges for prediabetes is between 5.7 to 6.4% for type II diabetes mellitus, it is between 7 to 9%.. For the current study, impaired range of Hba1c from 6.5 to 6.9% shall be consider as prediabetes

SECONDARY OUTCOMES:
Cohort 1- ( Pre-diabetes) To assess the effect of Investigational Product (IP) on blood sugar in Pre-diabetes as assessed by 2-hour plasma glucose level by Oral Glucose Tolerance Test | Screening visit (The same value will be considered for baseline) and Day 90.
  Oral glucose tolerance tests (OGTT) are used to measure how well the body can process a larger amount of sugar. If the blood sugar measured in the test is above a certain level, this could be a sign that sugar is not being absorbed enough by the body's cells. Diabetes or gestational diabetes might be at the root of this problem.As per American Diabetes Association, OGTT ranges for prediabetes individuals is 140 mg/ dL to 199 mg/dL and more than 200 mg/dl is considered as type II diabetes mellitus
Cohort 1- ( Pre-diabetes) To assess the effect of Investigational Product (IP) on blood sugar as assessed by Glucose metabolism as assessed by change in the HbA1c | Screening visit (The same value will be considered for baseline) and Day 90.
  HbA1c reference ranges for prediabetes is between 5.7 to 6.4% for type II diabetes mellitus, it is between 7 to 9%.. For the current study, impaired range of Hba1c from 6.5 to 6.9% is also being considered as prediabetes
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Pancreatic efficiency as assessed by the change in the fasting insulin | Day 0, Day 30, Day 60, Day 90
  Normal fasting insulin levels range between 5 and 15 μU/mL.
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Percentage change in body weight by weighing scale | Day 0, Day 30, Day 60, Day 90
  Obesity is a chronic condition characterized by an excess of body fat. It is a complex disorder of appetite regulation and energy metabolism controlled by specific biological factors. There is strong evidence to suggest that the risks of mortality and morbidity associated with obesity can be reduced with weight loss
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Change in central obesity as assessed by the change in the anthropometric index of waist-to-height ratio | Day 0, Day 30, Day 60, Day 90
  The waist circumference standardization should be conducted for the observer. Two measurements will be conducted for waist circumference and height. If the variance between the two readings is within ± 1 cm, a third measurement will be obtained. Similarly, two measurements will be taken for weight, and if the difference falls within ± 200 grams, a third measurement will be taken.
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Change in Fasting Blood Glucose (FBG) | Day 0, Day 30, Day 60, Day 90
  FBG measures blood sugar after an overnight fast. A fasting blood sugar level of 99 mg/dL or lower is normal, 100 to 125 mg/dL indicates prediabetes, and 126 mg/dL or higher indicates diabetes.
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Change in Quality of life as assessed by SF- 6Dv2TM Health Survey | Day 0, Day 30, Day 60, Day 90
  The quality of life will be assessed by SF- 6Dv2TM Health Survey. It is based on 6 health domains
  1. Physical functioning 2. Role functioning 3. Pain 4. Vitality 5. Social functioning 6. Mental health The quality of life of the participants will be analysed domain wise. Each domain will be rated from 0 to 5, 0 being worst and 5 being the best state.
Cohort 1 (Prediabetes) & Cohort 2 (T2DM): To assess the effect of Investigational product (IP) on Change in the Eating behavior as assessed by Three factor eating questionnaire - Revised 18 | Day 0, Day 30, Day 60, Day 90
  The raw scale scores are to be transformed to a 0-100 scale [((raw score - lowest possible raw score)/possible raw score range) × 100]. Higher scores in the respective scales are indicative of greater cognitive restraint, uncontrolled, or emotional eating
To assess the effect of Investigational product (IP) on:Lipid profile [total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides] | Screening visit (The same value will be considered for baseline) and Day 90.
  Insulin resistance, often associated with metabolic syndrome, can affect lipid metabolism. It may lead to increased levels of triglycerides and alterations in the balance of LDL and HDL cholesterol. High triglyceride levels are a common feature of metabolic syndrome. Excess calorie intake, especially from refined carbohydrates, can contribute to elevated triglycerides.

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Shourya clinic, Pune, Maharashta
  - Shri balaji Multispeciality hospital,, Thane, Maharashtra
  - Dr.Govinds Clinic,, Jaipur, Rajashthan
  - Upendra Medicare, Varanasi, Uttar Pradesh
  - Arihant Hospital, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No